CLINICAL TRIAL: NCT00899834
Title: Comprehensive Molecular Analysis of Tumor Samples Derived From Patients With Diffuse Brainstem Glioma - A Pilot Study
Brief Title: DNA Analysis of Tumor Tissue Samples From Patients With Diffuse Brain Stem Glioma
Status: Completed | Type: Observational
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: NBTP02-SJ
Record Dates: First submitted 2009-05-09; First posted 2009-05-12 (Estimated); Last update posted 2016-07-26 (Estimated); Status verified 2016-07

CONDITIONS: Brain Tumors; Central Nervous System Tumors
Keywords: adult brain stem glioma; childhood brain stem glioma
MeSH Terms: conditions — Brain Neoplasms; Central Nervous System Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — tumor and constitutional tissue samples from patients with diffuse brainstem glioma and other types of brainstem gliomas
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Tumor Samples: fresh-frozen and fixed tumor samples and correspondent normal tissue from patients affected with this tumor.(peripheral blood is applicable only to patients with focal brainstem gliomas and patients who undergo biopsy of a diffuse brainstem glioma at diagnosis)

SUMMARY:
This multi-institutional study will prospectively collect tumor and constitutional tissue samples from patients with diffuse brainstem glioma and other types of brainstem gliomas either during therapy or at autopsy to perform an extensive analysis of genetic and molecular abnormalities in these tumors.

DETAILED DESCRIPTION:
Since very little is known about the biology of diffuse brainstem glioma, the goal of this protocol is to undertake a systematic analysis of DNA abnormalities, and of RNA and protein expression in prospectively collected fresh-frozen and fixed tumor samples and correspondent normal tissue from patients affected with this tumor.

OBJECTIVES:

* Perform genome-wide analysis of DNA gains and losses and RNA expression in tumor samples and normal tissue from patients with diffuse brain stem glioma.
* Identify regions of genomic gain or loss using either array comparative genomic hybridization or single nucleotide polymorphism arrays.
* Investigate genome-wide expression patterns of RNA derived from tumor samples and normal tissue from these patients via Affymetrix gene expression profiling.
* Validate the results of the genome-wide analysis by conducting further evaluation of candidate genes or by investigating the expression of relevant gene products at the RNA and protein levels.
* Perform analysis of mutations in candidate tumor-suppressor genes and oncogenes (including whole genome sequencing studies) using direct sequence analysis of tumor DNA and confirm the tumor-specific nature of these mutations by analyzing the correspondent constitutional DNA.
* Confirm genomic gains or losses identified by means of fluorescence in situ hybridization (FISH) performed on tissue microarray using non-neoplastic brain tissue from each patient as control when available.
* Explore protein expression patterns identified by immunohistochemistry or western blot and compare them to normal brain stem tissue.
* To obtain a follow-up (questionnaire and/or telephone interview) after autopsy with parent(s), legal guardian(s), or family members of research participants in the United States to assess aspects associated with this procedure, including potential benefits and drawbacks

ELIGIBILITY:
Inclusion Criteria

* Patients of any age with clinical and radiologic diagnosis of diffuse brainstem glioma
* Patients with other high-grade gliomas originating in the brainstem
* Patients with focal gliomas (WHO grade I/II) of the brainstem
* Enrollment in the current version of the St. Jude Tissue Bank protocol for patients whose tissue samples were obtained at diagnosis and who received treatment at St. Jude Children's Research Hospital (SJCRH), or correspondent tissue banking consent for patients treated in other institutions if tissue was obtained prior to death (as applicable, depending on the standard of each institution)

Exclusion Criteria

* Patients with any type of infiltrative low-grade (WHO grade II) or high-grade glioma (WHO grade III and IV) originating outside the brainstem
* Patients harboring primary brainstem tumors with other histologic diagnoses (e.g., PNET)

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Fresh-frozen and fixed tumor samples and correspondent normal tissue from patients affected with this tumor (peripheral blood is applicable only to patients with focal brainstem gliomas and patients who undergo biopsy of a diffuse brainstem glioma at diagnosis)
Sampling Method: Non-Probability Sample
Enrollment: 81 (Actual)
Dates: Start 2006-06; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
DNA gains and losses and RNA expression in tumor samples and normal tissue | at autopsy
  Tissue samples will be obtained at autopsy.
Genome-wide expression patterns of RNA in tumor samples and normal tissue as assessed by Affymetrix gene expression profiling | at autopsy
  Tissue samples will be obtained at autopsy.
Validation of results of the genome-wide analysis | at autopsy
  Tissue samples will be obtained at autopsy.
Mutations in candidate tumor-suppressor genes and oncogenes as assessed by direct sequencing analysis of tumor DNA | at autopsy
  Tissue samples will be obtained at autopsy.
Confirmation of the tumor-specific nature of candidate tumor-suppressor gene and oncogene mutation as assessed by the correspondent constitutional DNA | at autopsy
  Tissue samples will be obtained at autopsy.
Confirmation of genomic gains or losses as assessed by fluorescence in situ hybridization (FISH) performed on tissue microarray (TMA) using non-neoplastic brain tissue | at autopsy
  Tissue samples will be obtained at autopsy.
Protein expression patterns as assessed by immunohistochemistry or western blot compared to normal brain stem tissue | at autopsy
  Tissue samples will be obtained at autopsy.

SECONDARY OUTCOMES:
Assess aspects associated with this procedure, including potential benefits and drawbacks | at autopsy
  Tissue samples will be obtained at autopsy.

CONTACTS AND LOCATIONS:
Overall Officials: Alberto Broniscer, MD, Principal Investigator — St. Jude Children's Research Hospital
Locations (3):
- United States (3):
  - Stanford University Medical Center, Palo Alto, California
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - Seattle Children's Hospital, Seattle, Washington

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols